CLINICAL TRIAL: NCT02699567
Title: CD36 Involvement on Fat Taste Perception and Fat Hedonic Value in Humans
Brief Title: CD36 and Human Fat Taste Perception
Acronym: FATYP
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: Monell Chemical Senses Center (Other)
Responsible Party: Principal Investigator, Marta Yanina Pepino de Gruev, Assistant Professor of Medicine, Washington University School of Medicine
Other Study IDs: 201011853
Record Dates: First submitted 2016-02-25; First posted 2016-03-04 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-02

CONDITIONS: Obesity
Keywords: taste perception; individual differences; fat; genetics
MeSH Terms: conditions — Obesity; Platelet Glycoprotein IV Deficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Extracted genomic DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Lean AA: Subjects with a BMI<=25 kg/m2 and carriers of a CD36 gene variation associated with low CD36 expression levels
  Interventions: Other: No intervention
- Obese AA: Subjects with a BMI>29.9 kg/m2 and carriers of a CD36 gene variation associated with low CD36 expression levels
  Interventions: Other: No intervention
- Lean GG: Subjects with a BMI<=25 kg/m2 and carriers of a CD36 gene variation associated with high CD36 expression levels
  Interventions: Other: No intervention
- Obese GG: Subjects with a BMI>29.9 kg/m2 and carriers of a CD36 gene variation associated with high CD36 expression levels
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
The purpose of this study is to determine the effect of common human variants in in taste related genes, such as CD36 gene, a putative fat taste receptor, affect fat taste perception.

DETAILED DESCRIPTION:
At present, the general agreement is that humans perceive five taste qualities: sweet, sour, bitter, salty and umami (the savory, meaty taste of some amino acids). It is believed that these qualities evolved to help us find nutrients (e.g. sweets, umami signaled calories) and avoid potential harmful substances (e.g. bitter signalized poison). Despite the fact that some fats, which can only be obtained through the diet, are essential for life, fat is not considered a basic taste; and, the issue of how fats are precisely sensed is unresolved. However, increasing evidence suggests that, in addition to smell and texture, taste plays an important role in fat perception. Putative fat taste receptor classes have been identified in animal models. One such receptor is the glycoprotein CD36, previously documented to be involved in trafficking and storage of fat. CD36 was recently found in rodents' and humans' taste buds. In rodents, CD36 deletion blunts specifically fat recognition. Although CD36 variants are frequent in humans, its role in humans' fat taste perception and preferences remains incompletely understood and will be the focus of the current proposal. The main goal of this study is to determine the effect of a common human variant in the CD36 gene on fat taste perception by using standardized sensory evaluation techniques. In addition, we will examine whether common variants in taste related genes (other than CD36) are associated with individual differences in the perception of flavors of milkshakes prepared with different amounts of fats.

ELIGIBILITY:
Inclusion Criteria:

* BMI >18-<25 kg/m2 or BMI>29.9 kg/m2.
* 21 to 50 years of age

Exclusion Criteria:

* Previous malabsorptive or restrictive gastrointestinal surgery
* Smoking
* Pregnancy or breastfeeding
* Diabetes
* Taking medication that might affect taste perception

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects will be men and women, 21 to 50 yrs of age of all races and ethnic groups. The two groups (i.e. groups with different CD36 genetic variants) will be matched as closely as possible in age, sex, body mass index and race distributions. Subject population will consist of lean subjects (BMI >18-<25 kg/m2) and subjects with obesity (BMI >29.9 kg/m2).
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2011-11; Primary Completion 2013-04 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Scores in the general labeled magnitude scale for fat flavor intensity | One to 12 weeks following screening
Scores in the hedonic general labeled magnitude scale for fat flavor hedonic value | One to 12 weeks following screening

SECONDARY OUTCOMES:
Number of participants who are PROP taster as assessed by sip and spit testing procedure of water with increasing PROP concentrations. | One to 12 weeks following screening

CONTACTS AND LOCATIONS:
Overall Officials: Marta Y Pepino de Gruev, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No